CLINICAL TRIAL: NCT04424368
Title: Creation and Evaluation of the Effectiveness of the Remote Monitoring System for Patients, Who Had Myocardial Infarction
Brief Title: Remote Monitoring System for Patients, Who Had Myocardial Infarction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ryazan State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 191119
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-08

CONDITIONS: Myocardial Infarction; Adherence, Patient
Keywords: myocardial infraction; the high level of potential adherence to treatment; polymorphism of genes; remote monitoring, prognosis
MeSH Terms: conditions — Myocardial Infarction; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The remote monitoring system (Experimental): A group of patients, who had myocardial infraction and who has a very high risk of developing an unfavorable prognosis, which are followed up in the local outpatient department according to existing clinical recommendations and using remote monitoring system.
  Interventions: Device: The remote monitoring system
- Clinical recommendations (No Intervention): A group of patients, who had myocardial infraction and who has a very high risk of developing an unfavorable prognosis, which are followed up in the local outpatient department according to existing clinical recommendations.

INTERVENTIONS:
Device: The remote monitoring system — Usage of remote monitoring system
  Arms: The remote monitoring system

SUMMARY:
one-centered, open, prospective, non-randomized, controlled clinical study will be aimed at creating remote monitoring system for patients' condition and the development of methodological approaches and its usage for conducting patients, who had myocardial infraction and who has a very high risk of developing an unfavorable outcome.

DETAILED DESCRIPTION:
The research will involve patients, who had myocardial infraction and who has the high level of potential adherence to treatment, which will be determined by the usage of Russian generic questionnaire for evaluation of compliance to drug therapy. At the end of a 12 month observation with the registration of unfavorable cardiovascular occasions (death from cardiovascular reasons, nonfatal myocardial infraction, cerebral stroke, necessity for repeated revascularization of the coronary arteries) based on the analysis of non-genetic and genetic factors (polymorphism of genes Thr174Met and Met235Thr in gene angiotensinogen, Arg389Gly and Ser49Gly in gene adrenoceptor beta 1, Ser447Ter in gene lipoprotein lipase and Leu28Pro in gene apolipoprotein E, Trp212Ter and G681A in gene cytochrome P450 family 2 subfamily C member 19) factors of unfavorable prognosis will be identified and considering which group of patients requires the use of remote monitoring system will be formed. From one group of patients we will form two comparable groups, one group will use this remote monitoring system and another will not. The effectiveness of the remote monitoring system will be evaluated after 6-month's observation based on the registration of the unfavorable cardiovascular occasions (death from cardiovascular reasons, nonfatal myocardial infraction, cerebral stroke, necessity for repeated revascularization of the coronary arteries, frequency of hospitalizations).

ELIGIBILITY:
Inclusion Criteria:

1. A significant diagnosis of myocardial infraction, confirmed by the level of biomarkers of myocardial necrosis in blood examination (troponin, creatine kinase-MV), electrocardiographic criteria, typical clinical presentation.
2. The high level of adherence to treatment
3. Signed informed agreement

Exclusion Criteria:

1. Active cancer or remission period less than 5 years;
2. Absolute contradictions to the prescription of beta-adrenergic blocking agents, angiotensin converting enzyme inhibitors, statins, antiaggregants.
3. Mental illnesses.
4. Alcohol and drug abuse
5. Patient's noncompliance, according to the researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-03 (Actual); Primary Completion 2021-12-03 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiovascular mortality | 12 months
  the number of deaths from cardiovascular causes
acute myocardial infarction | 12 months
  incidence of acute myocardial infarction
cerebral stroke | 12 months
  incidence of cerebral stroke
revascularization | 12 months
  frequency of repeated revascularization of coronary arteries
hospitalization | 12 months
  frequency of hospitalization about the progression of coronary heart disease

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Pereverzeva, MD, PhD, Principal Investigator — RyazSMU
Locations (1):
- RyazSMU, Ryazan, Russia

IPD SHARING:
Plan to Share IPD: No